CLINICAL TRIAL: NCT01042808
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy of ISENTRESS in Usual Practice
Brief Title: Isentress Re-examination Study (MK-0518-115)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0518-115; 2010_001 (Other: Merck)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infection; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: HIV-1 Infected patients treated with Isentress

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of Isentress through collecting the safety and efficacy information in usual practice according to the Re-examination Regulation for New Drugs.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Infected Adults
* Treated with Isentress 400 mg tablet within local label during the enrollment period

Exclusion Criteria:

* Contraindication to Isentress according to the local label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-1 Infected adults
Sampling Method: Probability Sample
Enrollment: 996 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with any adverse experience which occurs during treatment or within 14 days following cessation of treatment | up to 14 days after last treatment
Proportions of patients with HIV-1 RNA levels of less than 50 milliliter | 6 months after treatment +/- 2 weeks
Proportions of patients with HIV-1 RNA levels of less than 400 copies per milliliter | 6 months after treatment +/- 2 weeks
Change from baseline in CD4 cell count and overall efficacy evaluation by investigator (success, failure, or nonassessible) | 6 months after treatment +/- 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC